CLINICAL TRIAL: NCT07293845
Title: Can Nursing Students' Knowledge and Attitudes Toward Climate Change Be Strengthened for a Sustainable Future?: A Quasi-Experimental Study
Brief Title: Can Nursing Students' Knowledge and Attitudes Toward Climate Change
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Semanur Çelik Demiryürek, Research Assistant, Kastamonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 112425
Record Dates: First submitted 2025-11-13; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: University Student; Climate Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Module (Experimental): Training Module on Climate Change
  Interventions: Behavioral: Climate Module
- Standard Education (No Intervention): Standard Education

INTERVENTIONS:
Behavioral: Climate Module — Training Module on Climate Change
  Arms: Training Module

SUMMARY:
Climate change is a major global problem threatening individual health, public health, and health systems. Climate change poses a significant global threat to social and environmental health determinants, such as the disruption of food systems, the spread of climate-sensitive diseases, and the increased frequency and intensity of extreme weather events. The World Health Organization (WHO) estimates that climate change will cause approximately 250,000 additional deaths annually from malaria, diarrhea, malnutrition, and heat stress between 2030 and 2050. In this context, nursing students, as future healthcare providers, need to be prepared and knowledgeable about global warming, climate change and its impacts on health, climate change mitigation, adaptation and resilience, and the promotion of a healthy environment for a sustainable future. Therefore, the purpose of this study was to examine the effects of climate change education on nursing students' knowledge and attitudes regarding climate change and health.

DETAILED DESCRIPTION:
Climate change is a major global problem threatening individual health, public health, and health systems. Climate change poses a significant global threat to social and environmental health determinants, such as the disruption of food systems, the spread of climate-sensitive diseases, and the increased frequency and intensity of extreme weather events. The World Health Organization (WHO) estimates that climate change will cause approximately 250,000 additional deaths annually from malaria, diarrhea, malnutrition, and heat stress between 2030 and 2050. Climate change leads to increased mortality and illness due to extreme weather events such as heat waves, storms, and floods; increases in the frequency and intensity of food-borne, water-borne, and vector-borne infectious diseases; exacerbations of chronic diseases; and increases in mental health problems. Consequently, it negatively impacts individual health physically, mentally, and socially. Due to the increasingly negative impacts of climate change on human health, nurses can serve as expert resources for patients, community members, and policymakers. However, nurses need to be well-equipped and highly aware of this issue. In this context, it is emphasized that nurses' climate-related competencies should be enhanced both today and in the future, starting with the educational process and developing independent practices rather than topics covered in existing courses. In this context, nursing students, as future healthcare providers, need to be prepared and knowledgeable about global warming, climate change and its impacts on health, climate change mitigation, adaptation and resilience, and the promotion of a healthy environment for a sustainable future. Therefore, the purpose of this study was to examine the effects of climate change education on nursing students' knowledge and attitudes regarding climate change and health.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th-year nursing student
* Voluntarily participating

Exclusion Criteria:

* Having any situation that would prevent communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Climate, Health, and Nursing Tool | 8 weeks
  The Climate, Health, and Nursing Tool (CHANT) was developed by Schenk and colleagues (2016). The Turkish validity and reliability study was conducted by Yalçın and Aktaş, and the scale can be used to assess awareness of climate change as well as knowledge and attitudes regarding the climate-health relationship. The scale consists of 48 items and five subdimensions: knowledge, awareness, motivation, concern, and behaviors. There is no total scale score; instead, evaluations are based on subdimension scores. In the validity and reliability analysis, the Cronbach's alpha value for the overall scale was reported as 0.93; for the knowledge subdimension 0.78, for awareness 0.97, for motivation 0.89, for concern 0.95, and for behaviors 0.94.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ARABACI, pHD, Study Director — Kastamonu University
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Result] Colak M, Dogan R, Dogan S. Effect of Climate Change and Health Course on Global Warming Knowledge and Attitudes, Environmental Literacy, and Eco-Anxiety Level of Nursing Students: A Quasi-Experimental Study. Public Health Nurs. 2025 May-Jun;42(3):1315-1324. doi: 10.1111/phn.13536. Epub 2025 Jan 17. PMID 39822057
- See also: World Health Organization (WHO) — https://www.who.int/news-room/fact-sheets/detail/climate-change-and-health